CLINICAL TRIAL: NCT05484622
Title: A Phase 1, Safety Lead-In and Randomized, Open-label, Perioperative Study of Vorasidenib in Combination With Pembrolizumab in Subjects With Recurrent or Progressive IDH-1 Mutant Glioma
Brief Title: Study of Vorasidenib and Pembrolizumab Combination in Recurrent or Progressive IDH-1 Mutant Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95032-005; MK-3475-B39 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-07-21; First posted 2022-08-02 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Astrocytoma; Oligodendroglioma
Keywords: Vorasidenib; AG-881; Pembrolizumab; IDH-1; Astrocytoma; Oligodendroglioma; Enchancing; Non-enchancing
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — vorasidenib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Sequential design for safety lead-in and randomized perioperative phases, parallel design within randomized perioperative phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Lead-In Phase: Vorasidenib + Pembrolizumab (Experimental): Participants will receive vorasidenib orally, once daily (QD) in combination with pembrolizumab 200 mg intravenous (IV) infusion, once every 3 weeks (Q3W) in each 21-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Interventions: Drug: Vorasidenib; Drug: Pembrolizumab
- Randomized Perioperative Phase: Vorasidenib + Pembrolizumab (Experimental): Participants will receive vorasidenib recommended combination dose (RCD) determined in the Safety Lead-in phase, orally, QD from Day 1 to 28 in combination with pembrolizumab 200 mg IV infusion, Q3W on Days 1 and 22 of a 28-day cycle prior to surgery.
  Interventions: Drug: Vorasidenib; Drug: Pembrolizumab
- Randomized Perioperative Phase: Vorasidenib Only (Experimental): Participants will receive vorasidenib orally, QD from Day 1 to 28 of a 28-day cycle prior to surgery.
  Interventions: Drug: Vorasidenib
- Randomized Perioperative Phase: Untreated Control Group (No Intervention): Participants will not receive any treatment prior to surgery.

INTERVENTIONS:
Drug: Vorasidenib — Administered orally as tablets.
  Other Names: S095032; AG-881
  Arms: Randomized Perioperative Phase: Vorasidenib + Pembrolizumab; Randomized Perioperative Phase: Vorasidenib Only; Safety Lead-In Phase: Vorasidenib + Pembrolizumab
Drug: Pembrolizumab — Administered as IV infusion.
  Other Names: MK-3475; KEYTRUDA®; KEYNOTE-B39; MK-3475-B39
  Arms: Randomized Perioperative Phase: Vorasidenib + Pembrolizumab; Safety Lead-In Phase: Vorasidenib + Pembrolizumab

SUMMARY:
Vorasidenib in combination with pembrolizumab in participants with recurrent or progressive isocitrate dehydrogenase-1 (IDH-1) mutant Glioma.

DETAILED DESCRIPTION:
The study is divided into 2 phases, a Safety Lead-In phase and a randomized perioperative phase. In the Safety Lead-In Phase, the recommended combination dose (RCD) of vorasidenib will be determined. In the Randomized Perioperative Phase, the Lymphocytes infiltration in tumors will be evaluated following pre-surgical treatment with vorasidenib and pembrolizumab combination, compared to untreated control tumors. Prior to surgery, participants will be randomized to receive vorasidenib at the RCD in combination with pembrolizumab, or vorasidenib only, or no treatment (untreated control group). Following surgery, participants will have the option to receive treatment with vorasidenib in combination with pembrolizumab in 21-day cycles.

Study treatment will be administered until participant experiences unacceptable toxicity, disease progression, or other discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

1. Have Karnofsky Performance Status (KPS) of ≥ 70%.
2. Have expected survival of ≥ 3 months.
3. Have histologically confirmed Grade 2 or Grade 3 glioma (per the 2016 or 2021 World Health Organization [WHO] Classification of Tumors of the central nervous system)
4. Have:

   1. Documented IDH1-R132H gene mutation; and
   2. For Astrocytomas: Absence of 1p19q co-deletion (i.e., exclusion of combined whole-arm deletions of 1p and 19q) and/or documented loss of nuclear ATRX expression or ATRX mutation by local testing. For Oligodendrogliomas: Presence of 1p19q co-deletion (i.e., combined whole-arm deletions of 1p and 19q) by local testing.
5. Have measurable, magnetic resonance imaging (MRI)-evaluable, unequivocal contrast enhancing disease as determined by institutional radiologist/Investigator at Screening on either 2D T1 post-contrast weighted images or 3D T1 post-contrast weighted images. Per mRANO criteria, measurable lesion is defined as at least 1 enhancing lesion measuring ≥ 1 cm x ≥ 1 cm. OR (in the absence of measurable enhancing disease) measurable, MRI-evaluable, unequivocal non enhancing disease as determined by institutional radiologist/Investigator at Screening on either 2D or 3D T2-weighted image or FLAIR. Per RANO 2.0 criteria, measurable lesion is defined as at least 1 non enhancing lesion measuring ≥ 1 cm × ≥ 1 cm.
6. Have recurrent or progressive disease and received prior treatment with chemotherapy, radiation, or both.
7. Surgical resection is indicated for treatment, but surgery is not urgently indicated (e.g., for whom surgery within the next 6-9 weeks is appropriate). (NOTE: This criterion only applies to participants enrolled in the perioperative phase of the study. Participants in the Safety Lead-In should not require surgery).

Exclusion Criteria:

1. Have received prior systemic anti-cancer therapy within 1 month of the first dose of IMP, radiation within 12 months of the first dose of IMP, or an investigational agent < 14 days prior to the first dose of IMP. In addition, the first dose of IMP should not occur before a period of ≥ 5 half-lives of the investigational agent has elapsed.
2. Have received 2 or more courses of radiation.
3. Have received any prior treatment with an isocitrate dehydrogenase (IDH) inhibitor; anti-programmed cell death 1 (PD1), anti-programmed cell death ligand 1 (PD-L1), or anti-PD-ligand 2 (L2) agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137); any other checkpoint inhibitor; bevacizumab; or any prior vaccine therapy.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Phase: Percentage of Participants With Dose-limiting Toxicities (DLTs) | First 21 days of dosing (Cycle 1) in safety lead-in phase
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | approximately up to 19 months
Percentage of Tumor-infiltrating Lymphocyte (TIL) Cells in Surgically Resected Tumors Following Treatment With Vorasidenib + Pembrolizumab Compared to Untreated Control Tumors | approximately 2 months
  TIL is defined as the percentage of tumor-infiltrating lymphocyte cells on a logarithmic scale.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 55 months
  Overall survival is defined as the time from the date of first dose (in Safety Lead-in) or first postoperative dose (in randomized perioperative phase) to the date of death due to any cause.
AUC: Area Under the Plasma Concentration-Time Curve of Vorasidenib | approximately 16 months
Cmax: Maximum Observed Plasma Concentration of Vorasidenib | approximately 16 months
Concentration of 2-hydroxygluarate (2-HG) in Surgically Resected Tumors | approximately 2 months
Concentration of Vorasidenib in Surgically Resected Tumors | approximately 2 months
Clinical Activity Associated With Vorasidenib in Combination With Pembrolizumab According to Modified Response Assessment in Neuro-oncology (mRANO) Criteria | Up to approximately 16 months
Time to response | Up to approximately 55 months
  Defined as the time from the date of first dose (in Safety Lead-In) or the date of first postoperative dose (in randomized perioperative phase) to the date of first documented objective response as assessed by the Investigator per Modified Response Assessment in Neuro-oncology (mRANO) criteria.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles (Site: 840113), Los Angeles, California
  - University of California, San Francisco (Site: 840149), San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Miami (Site: 840129), Miami, Florida
  - Northwestern University (Site: 840123), Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital (Site: 840104), Boston, Massachusetts
  - Dana-Farber Cancer Institute (Site: 840139), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center (Site: 840117), New York, New York
  - Duke University (Site: 840110), Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Mayo Clinic Florida, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center (Site: 840102), Houston, Texas
  - University of Utah, Huntsman Cancer Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * Used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * Sponsored by Servier
  * With a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Wen P, Peters K, de la Fuente M, Mellinghoff I, Arrillaga-Romany I, Kumthekar P, Clarke J, Puduvalli V, de Groot J, Zhang J, Chisamore M, Abshire M, Mahboub P, Hassan I, Knipstein J, Cloughesy T. Phase 1 Safety Lead-in and Randomized Open-label Perioperative Study of Vorasidenib Combined with Pembrolizumab in Recurrent or Progressive Enhancing IDH1-mutant Astrocytomas: Safety Lead-in Results. Neuro Oncol. 2023 Nov 10;25(Supplement_5):V65. doi: https://doi.org/10.1093/neuonc/noad179.0254